CLINICAL TRIAL: NCT01253876
Title: Effect of Soymilk Replacement on Anthropometric and Blood Pressure Value
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Other Study IDs: Soy milk weight blood pressure
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-03

CONDITIONS: Weight; Waist; Systolic Blood Pressure; Diastolic Blood Pressure
MeSH Terms: conditions — Body Weight | interventions — Soy Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soy milk (Experimental)
  Interventions: Dietary Supplement: soy milk, Caw's milk
- Caw's milk (Experimental)
  Interventions: Dietary Supplement: soy milk, Caw's milk

INTERVENTIONS:
Dietary Supplement: soy milk, Caw's milk

SUMMARY:
Soymilk components such as isoflavones, essential fatty acids, phytoesterols, good fats, inositols might have beneficial effects on weight control and blood pressure management. Most studies in this regard have been conducted on postmenopausal or premenopausal women and there are few studies on female youths. Therefore, we are going to determine the effects of soy consumption on the weight, waist circumference and blood pressure in overweight and obese female youths. This was a cross-over randomized clinical trial which was conducted in 2010 in Isfahan on overweight or obese young female youths. After three weeks run-in, females were randomly assigned to consume a diet containing caw's milk or a diet in which only one glass of soy milk was substituted; each one for six weeks. Random sequencing generated in SPSS was used for allocating females in different group randomly. Patients were not blinded because they had to use soy milk in one period of trial and use caw's milk in another period.

ELIGIBILITY:
Inclusion Criteria:Being in the age range of 18 to 30 and having body mass index more than 30 kg/m2 were the inclusion criteria.

-

Exclusion Criteria:Having allergy to soy product or caw's milk and not consuming the soy milk or caw's milk, incidence of chronic or acute diseases which make patients not to follow the research protocol or beginning to consume the medications were the exclusion criteria.

-

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Iran